CLINICAL TRIAL: NCT02289794
Title: Evaluation of a Candidate Vaccine Against Uropathogenic Escherichia Coli in Women With a Clinical History of Recurrent Urinary Tract Infection
Brief Title: Vaccine Against Escherichia Coli Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoVaxyn AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GVXN EC-4V; 2013DR1205 (Other: swissmedic)
Record Dates: First submitted 2014-11-03; First posted 2014-11-13 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: E.Coli Infections
Keywords: Bioconjugate vaccine; Urinary tract infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E.coli bioconjugate vaccine (Active Comparator): E.coli bioconjugate vaccine in saline buffer
  Interventions: Biological: E.coli bioconjugate vaccine
- Placebo (Placebo Comparator): Saline buffer
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: E.coli bioconjugate vaccine — Single dose, intramuscular injection (0.5 mL)
  Other Names: EcoXyn-4V
  Arms: E.coli bioconjugate vaccine
Biological: Placebo — Single dose, intramuscular injection (0.5 mL)
  Arms: Placebo

SUMMARY:
This Phase I multi-center placebo controlled study is conducted in healthy women with a history of recurrent urinary tract infections (UTI) aged between 18 and 70 years.

DETAILED DESCRIPTION:
GlycoVaxyn is a Swiss company that has developed a multivalent bioconjugate vaccine for the prevention of E.coli-infections. Cystitis is the most common UTI, however kidney infections or bacteremia are possible. The E. coli bacterium is responsible for 85 % of all UTIs.

The objectives of this trial are to assess the safety and ability to elicit an immune response of the candidate vaccine as well as the effectiveness of the vaccine in the reduction in UTIs .

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects with a history of recurrent UTI, which is defined as: ≥ 3 UTI independent episodes in the previous 12 months or ≥ 2 UTI episodes in the last 6 months. At least one UTI during the last 5 years was caused by E. coli (as single pathogen or part of polymicrobial infection) and was culture-confirmed and documented
2. Age ≥ 18 and ≤ 70 years
3. Subjects should be in a healthy state without ongoing or suspected symptomatic UTI at the screening visit and at injection day (V2)
4. General good health, without clinically significant medical history, physical examination findings or clinical laboratory abnormalities per clinical judgment of the investigator
5. Willingness to participate in the study after all aspects of the protocol have been explained and fully understood, and written informed consent form obtained

Exclusion Criteria:

1. History of more than 10 recurrent UTIs in the year before the screening visit
2. Use of any short-term urinary catheter within 7 days prior to screening
3. Use of any permanent catheter within 30 days prior to screening
4. History of any unresolved urinary tract diseases/abnormalities
5. Evidence of impaired immune function
6. Significant cardiovascular, liver, renal diseases and/or insufficiency
7. Uncontrolled diabetes mellitus
8. Significant abnormalities in screening results for hematology, serum chemistry or urinalysis
9. Positive test for HIV, and/or evidence of HBV or HCV
10. BMI >34
11. Previous immune stimulatory therapy for UTI prevention (such as Urovaxom®, Strovac® or Urovac®) in the last 3 months, or planned use during the study period
12. Current use of any medication known to affect immune function (e.g. corticosteroids ≥0.5 mg/kg Body weight/day)
13. Use of UTI-related vaginal estrogen treatment newly started less than 6 months before injection and continuing during the study or planned start during the active study period
14. Use of any antibiotic therapy within 1 week preceding injection
15. Planned use of post-coital antibiotics for UTI prevention during study period
16. Any vaccination planned within 30 days before and 30 days after injection
17. Participation in other clinical trials in the 60 days preceding enrolment and for the duration of the study
18. Previous treatment with immunoglobulins or blood products in the 3 months preceding the injection
19. Known hypersensitivity to any component of the vaccine
20. Presence of a significant medical or psychiatric condition that in the opinion of the investigator precludes participation in the study
21. Acute illness at the time of injection
22. Women of child bearing potential who either have a positive pregnancy test or refuse to use an effective contraception
23. Women who are lactating at any time throughout the study period
24. Subjects with an elective surgical intervention, planned during the study period
25. Any other significant finding that in the opinion of the Investigator would increase the risk of having an adverse outcome from participating in the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing an adverse events | 30 days
  Occurrence, intensity, relationship and duration of solicited and unsolicited adverse events (AE) and serious adverse events (SAE) post injection of candidate vaccine compared to the placebo group

SECONDARY OUTCOMES:
Comparison of E.coli vaccine-specific serotypes antibody concentrations in serum at different timepoints | 30 days and 9 months
  Evaluation of IgG Response of candidate vaccine between baseline (D1) and post injection (D30 and D270)

OTHER OUTCOMES:
Reduction of UTI episodes caused by E.coli vaccine-specific serotypes | 9 months
  Comparison of the number of symptomatic UTI episodes caused by E. coli vaccine-serotypes between the two arms, injected with candidate-vaccine or placebo during the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Gambillara, PhD, Study Director — GlycoVaxyn AG
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huttner A, Hatz C, van den Dobbelsteen G, Abbanat D, Hornacek A, Frolich R, Dreyer AM, Martin P, Davies T, Fae K, van den Nieuwenhof I, Thoelen S, de Valliere S, Kuhn A, Bernasconi E, Viereck V, Kavvadias T, Kling K, Ryu G, Hulder T, Groger S, Scheiner D, Alaimo C, Harbarth S, Poolman J, Fonck VG. Safety, immunogenicity, and preliminary clinical efficacy of a vaccine against extraintestinal pathogenic Escherichia coli in women with a history of recurrent urinary tract infection: a randomised, single-blind, placebo-controlled phase 1b trial. Lancet Infect Dis. 2017 May;17(5):528-537. doi: 10.1016/S1473-3099(17)30108-1. Epub 2017 Feb 24. PMID 28238601